CLINICAL TRIAL: NCT06725550
Title: Integrative Medicine in Pain Management in Sickle Cell Disease: Assessing the Clinical Efficacy and Neurobiological Impact With Acupuncture, 2.0
Brief Title: Integrative Medicine in Pain Management in Sickle Cell Disease, 2.0
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Ying Wang, Assistant Professor of Anesthesia, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 25633
Record Dates: First submitted 2024-12-05; First posted 2024-12-10 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Sickle Cell Disease; Pain; Acupuncture; Quantitative Sensory Testing; Magnetic Resonance Imaging; Circulating Biomarkers; Electroencephalography; Functional Near-infrared Spectroscopy
Keywords: Sickle cell disease; Pain; Acupuncture; Quantitative Sensory Testing; Magnetic Resonance Imaging; Circulating Biomarkers; Electroencephalography; Functional Near-infrared Spectroscopy
MeSH Terms: conditions — Anemia, Sickle Cell; Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- Needling Acupuncture - 5 weeks (Experimental): Needling acupuncture treatment will last 30 minutes per session and will be administered two times per week for 5 weeks. Each subject will receive one course of treatment which contains 10 treatment sessions.
  Interventions: Device: needling acupuncture
- Laser Acupuncture - 5 weeks (Experimental): Laser acupuncture treatment will also last 30 minutes per session and will be administered two times per week for 5 weeks. Each subject will receive one course of laser acupuncture treatment which contains 10 treatment sessions.
  Interventions: Device: laser acupuncture
- Needling Acupuncture - 12 weeks (Experimental): Needling acupuncture treatment will last 30 minutes per session and will be administered once per week for 12 weeks. Each subject will receive one course of treatment which contains 12 treatment sessions.
  Interventions: Device: needling acupuncture
- Laser Acupuncture - 12 weeks (Experimental): Laser acupuncture treatment will also last 30 minutes per session and will be administered once per week for 12 weeks. Each subject will receive one course of laser acupuncture treatment which contains 12 treatment sessions.
  Interventions: Device: laser acupuncture

INTERVENTIONS:
Device: needling acupuncture — Acupuncture treatment will both main and supplementary acupoints. Main points include GB30; ST36; LI11- LI4, GB34-SP6; LR3, SP10, DU24, DU20, Yin Tang, Ear Shen Men which are chosen based on the unique clinical features of sickle pain. The remaining individualized acupoints will be selected and manipulated with manual acupuncture with appropriate needling techniques based on the individual "Syndrome" ("reinforce" or "reduce" or "Non reinforce or reduce") that is determined by TCM diagnosis.
  Arms: Needling Acupuncture - 12 weeks; Needling Acupuncture - 5 weeks
Device: laser acupuncture — Laser acupuncture device VitaLaser 650 (Lhasa OMS, Weymouth, MA or similar) will be positioned 1-2cm over all of the same acupoints used in verum acupuncture treatment above. No palpation is administered prior to positioning the device and there is no physical contact between device and skin.
  Arms: Laser Acupuncture - 12 weeks; Laser Acupuncture - 5 weeks

SUMMARY:
The proposed research is to determine the clinical efficacy and neurobiological mechanisms of acupuncture analgesia in patients with sickle cell disease.

DETAILED DESCRIPTION:
This study will help the investigators to learn whether acupuncture, which is a non-opioid alternative pain management approach, can help to manage pain in patients with sickle cell disease and the underlying mechanisms. Acupuncture involves inserting very fine needles through the skin at specific points on the body to different depths. Acupuncture may help relieve pain and it is used for a wide range of pain conditions. Participation in this study will include 14 study visits over around 6-8 weeks and 12 months follow-up visits. This is a randomized study, which means subjects are randomly assigned to one of two groups. During the study visits: 1) Subjects will be randomized to 10 sessions with either traditional acupuncture (very fine acupuncture needles will be inserted into the skin) or laser acupuncture without needles (a laser acupuncture device will be used and there will be no physical contact between the device and subject's skin) and each session will last for 30 minutes, 2) Subjects will answer questions about their personal and health related information for assessing health condition during the in-person and follow-up study visits, 3) Investigators will perform quantitative sensory testing (QST) before and after the acupuncture sessions on the surface of selected testing areas in subjects to assess the somatosensory functionality, 4) Investigators will record brain signals before and after acupuncture sessions using magnetic resonance imaging (MRI)-an imaging tool to analyze brain structural and functional features and metabolites profile, functional near-infrared spectroscopy (fNIRS)-an imaging tool to examine the brain hemodynamic activity, and electroencephalography (EEG) -an imaging tool used to detect the brain electrical activity, 5) Subjects will receive evoked pain stimuli on the left gastrocnemius muscle during MRI, fNIRS and EEG, 6) Female subjects will take a urine pregnancy test during the screening visit as well as before each behavioral and MRI visit, 7) Investigators will collect an inner eyelid image collection for examining the hemoglobin level and 8) subjects will have two blood draws before and after the entire acupuncture sessions for regular blood examination and circulating biomarkers' analyses. Some details regarding the interventions are purposefully omitted at this time to preserve scientific integrity. They will be included after the trial is complete.

ELIGIBILITY:
Inclusion Criteria:

* Any gender
* 14-17 (Adolescents) and 18-80 (Adults) years old
* Right-handed
* Either outpatient or inpatient or status changing between each other
* Have been diagnosed with SCD (includes but not limited to SS, SC or other type) and experiencing chronic pain in the past 6 months or vaso-occlusive crisis (VOC) in the past 12 months.
* Analgesic therapy prescribed by primary hematologists (or physicians for emergency or primary care) including pain-relieving medications (e.g. Morphine, coderin, Fentanyl, Oxycodone), Hydroxyurea (e.g. Droxia, Hydrea, Siklos), L-glutamine oral powder (Endari), Crizanlizumab (Adakveo), Voxelotor (Oxbryta), and/or other palliative treatment allowed, not required.
* Willing to limit the current and the introduction of any new medications or treatment modalities for control of pain symptoms during the study visits.
* Able to travel to the study site for participating scheduled visits (questionnaires, QST, EEG and MRI) and receive acupuncture treatments up to two times weekly for 5 weeks as scheduled.
* We will recruit without regard to ethnicity, however, due to the genetic nature of SCD, subjects will primarily be African-American or of African descent, although there are individuals with SCD who come from Hispanic, southern European, Middle Eastern, or Asian Indian backgrounds. The ethnic distribution in our prior studies is 95% Black/African American with 5% Hispanic or Latino (of any race). As these are minority groups many individuals may be from lower income situations.
* Fluent in English and capable of giving written informed consent.

Exclusion Criteria:

* Subjects with Covid-19 suspicion or confirmation
* Recent/ongoing alternative pain management with acupuncture or acupuncture-related techniques within the last 6-months.
* Presence of a known coagulation abnormality: Thrombocytopenia (mild thrombocytopenia with a platelets range of 51,000-100,000/ul will be further evaluated for inclusion consideration), or bleeding diathesis that may preclude the safe use of acupuncture.
* Presence of a concurrent autoimmune or inflammatory disease such as rheumatoid arthritis, systemic lupus erythematosus, inflammatory bowel disease, etc. that causes pain or any other chronic pain condition with pain greater than sickle pain.
* Diseases/conditions history includes but not limited to:

  * head injury with substantial loss of consciousness
  * peripheral neuropathy of known cause that interferes with activities of daily living
  * known non-SCD related Severe psychiatric illnesses (e.g. current schizophrenia, major depression with suicidal ideation).
  * significant visual, motor, or auditory impairment that would interfere with ability to perform study visits-related activities
* Medication:

Recent (30 days) initiation or dose adjustment of stimulant medications, such as those used to treat ADD/ADHD (e.g., amphetamine/dextroamphetamine [Adderall®], methylphenidate, dextroamphetamine), or the fatigue associated with sleep apnea or shift work (e.g., modafinil).

* Contraindications to MRI scans includes but are not limited to: surgical clips, surgical staples, metal implants, cardiac rhythmic disorders, seizure disorders, and certain metallic dental material will not be scheduled for MRI visits.
* History vascular surgery in lower limbs or current lower limb vascular dysfunction will not receive conditioned pressure pain stimuli in the lower limb.
* Subjects with Worker's Compensation, Workman's Compensation, civil litigation or disability claims pertinent to the subject's sickle disease; current involvement in out-of-court settlements for claims pertinent to the subject's sickle disease; or currently receiving monetary compensation as a result of any of the above.
* Participation of other studies: Concurrent participation in other therapeutic trials with overlapping research purposes.
* Pregnant or nursing.

Ages: 14 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-08-25 (Actual); Primary Completion 2029-08-31 (Estimated); Study Completion 2030-08-30 (Estimated)

PRIMARY OUTCOMES:
Functional brain connectivity characteristics | changes brain connectivity features from baseline to post-treatment time point (approximately 5 weeks interval)
  Characteristics of functional brain activity will be studied using fMRI.
Somatosensory function | changes of quantitative sensory testing scores from baseline to post-treatment time point (approximately 5 weeks interval)
  Somatosensory functionality will be examined using a board tests of which is a reliable and reproducible approach in pain research.

SECONDARY OUTCOMES:
Brain metabolites characteristics | changes of brain metabolites levels from baseline to post-treatment time point (approximately 5 weeks interval)
  Characteristics of brain metabolites will be studied using 1H-MRS.
painDETECT Questionnaire | changes of painDETECT scores from baseline to post-treatment time point (approximately 5 weeks interval)
  This is 4-component questionnaires that address the location, intensity, quality of pain symptoms. painDETECT is a nine-item questionnaire that consists of seven sensory symptom items for pain that are graded from 0= never to 5= strongly, one temporal item on pain-course pattern graded -1 to +1, and one spatial item on pain radiation graded 0 for no radiation or +2 for radiating pain.
Brief Pain Inventory (BPI) Questionnaire | changes of BPI scores from baseline to post-treatment time point (approximately 5 weeks interval)
  A simplified BPI is used to assess the severity of pain, interference of pain on daily function, location of pain, pain medications and amount of pain relief using the rating from 0= no pain/relief/interference to 10= worst pain imaginable/complete relief/completely interferes in the past 24 hours or the past week.
Nociplastic Pain Questionnaire | changes of nociplastic scores from baseline to post-treatment time point (approximately 5 weeks interval)
  A customized questionnaire that is used to examine the locations (Yes/No) and severity of the pain interference (no problem-slight-moderate--severe) for understanding the level of nociplastic pain in the past 7 days. Widespread Pain Index and Symptom Severity will be scored from 0 to 10. Higher score connotes higher severity of nociplastic pain.
Hospital Anxiety and Depression Scale (HADS) Questionnaire | changes of HADS scores from baseline to post-treatment time point (approximately 5 weeks interval)
  HADS is used to determine the levels of anxiety and depression that a person is experiencing in the past one week. The HADS is a fourteen-item scale that generates: Seven of the items relate to anxiety and seven relate to depression. Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 and 21 for either anxiety or depression.
Psychological Screening Questionnaires (PHQ-9) | changes of PHQ-9 scores from baseline to post-treatment time point (approximately 5 weeks interval)
  PHQ-9 is used to assess the mental health conditions in the past two weeks. Total scores of 5, 10, 15, and 20 represent cut points for mild, moderate, moderately severe, and severe depression, respectively.
Patient-Reported Outcomes Measurement Information System (PROMIS)-29 Questionnaire | changes of PROMIS-29 scores from baseline to post-treatment time point (approximately 5 weeks interval)
  The PROMIS-29 has seven health domains (physical function, fatigue, pain interference, depressive symptoms, anxiety, ability to participate in social roles and activities, and sleep disturbance) with customized 29-item questions and a single 4-20 numeric rating for each question.
Multidimensional Fatigue Inventory (MFI) Questionnaire | changes of MFI scores from baseline to post-treatment time point (approximately 5 weeks interval)
  MFI is a 20-item self-report instrument designed to measure fatigue with five dimensions including General Fatigue, Physical Fatigue, Mental Fatigue, Reduced Motivation and Reduced Activity. Subscale scores (range 4-20) are calculated as the sum of item ratings and a total fatigue score (range 20-100) is calculated as the sum of subscale scores. Higher scores indicate a higher level of fatigue.
Pittsburgh Sleep Quality Index (PSQI) Questionnaire | changes of PSQI scores from baseline to post-treatment time point (approximately 5 weeks interval)
  The PSQI is a 19-item, self-rated questionnaire designed to measure sleep quality and disturbance over the past month in clinical populations. The sleep component scores are summed to yield a total score ranging from 0 to 21 with the higher total score (referred to as global score) indicating worse sleep quality.
Adult Sickle Cell Quality Measure (ASCQ-ME) Questionnaire | changes of pain-related quality of life scores from baseline to post-treatment time point (approximately 5 weeks interval), as well as monthly follow-up visits till the 12th month of last in-person visit.
  ASCQ-Me contains both questionnaires of pain episodes frequency, severity, and the pain impact that can comprehensively examine the disease severity and impact in pain, stiffness, sleep, social function in patients with SCD. Scores for ASCQ-Me impact scales range from 0 to 100, with a standardized SCD population mean of 50 (SD, 10), where lower scores connote worse disease impact.
Pediatric Quality of Life Inventory (PedsQL, both pediatric and adult versions) Questionnaire | changes of pain-related quality of life scores from baseline to post-treatment time point (approximately 5 weeks interval), as well as monthly follow-up visits till the 12th month of last in-person visit.
  The PedsQL is a self-report and parent-report measure assessing the quality of life in a variety of domains including physical, emotional, social, and school. Items are reverse-scored and transformed to a 0-100 scale where higher scores indicate better quality of life.

OTHER OUTCOMES:
Circulating biomarkers' profile and levels | changes of circulating biomarkers levels from baseline to post-treatment time point (approximately 5 weeks interval)
  Circulating biomarkers' expression profile and quantitative level of each targeted biomarker in blood samples will be examined using proteomics, multiplex assays, ELISA and etc.
Blood hemoglobin level | changes of blood hemoglobin level from baseline to post-treatment time point (approximately 5 weeks interval)
  Blood hemoglobin level will be assessed by both regular blood sample analysis and a patented algorithm of spectral super-resolution spectroscopy technique using a software installed smartphone through the participants' inner eyelid.
Brain hemodynamic activity | changes of brain hemodynamic activity from baseline to post-treatment time point (approximately 5 weeks interval)
  Brain hemodynamic activity will be recorded and examined by functional near-infrared spectroscopy.
Brain structural characteristics | changes of brain structural characteristics from baseline to post-treatment time point (approximately 5 weeks interval)
  Brain structural features will also be examined using MRI.
brain electrophysiological characteristics: EEG power in alpha band | changes of alpha band from baseline to post-treatment time point (approximately 5 weeks interval)
  Brain electrophysiological signals will be recorded and examined by EEG. EEG power in alpha band will be analyzed using Matlab, EEGLab or other computer software designed for EEG data.
brain electrophysiological characteristics: EEG power in theta band | changes of theta band from baseline to post-treatment time point (approximately 5 weeks interval)
  Brain electrophysiological signals will be recorded and examined by EEG. EEG power in theta band will be analyzed using Matlab, EEGLab or other computer software designed for EEG data.
brain electrophysiological characteristics: EEG power in beta band | changes of beta band from baseline to post-treatment time point (approximately 5 weeks interval)
  Brain electrophysiological signals will be recorded and examined by EEG. EEG power in beta band will be analyzed using Matlab, EEGLab or other computer software designed for EEG data.
brain electrophysiological characteristics: EEG power in delta band | changes of delta band from baseline to post-treatment time point (approximately 5 weeks interval)
  Brain electrophysiological signals will be recorded and examined by EEG. EEG power in delta band will be analyzed using Matlab, EEGLab or other computer software designed for EEG data.

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University School of Medicine, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang Y, Hardy SJ, Ichesco E, Zhang P, Harris RE, Darbari DS. Alteration of grey matter volume is associated with pain and quality of life in children with sickle cell disease. Transl Res. 2022 Feb;240:17-25. doi: 10.1016/j.trsl.2021.08.004. Epub 2021 Aug 19. PMID 34418575
- [Result] TJ Barrett, A Pucka, B Reyes, SA Jacob, ARW O'Brien, RE Harris, SE Harte, Y Wang*. Acupuncture Alleviates Pain and Improves Quality of Life in Patients with Sickle Cell Disease. Blood. (2022);140 (Supplement 1):5444-5445. (https://doi.org/10.1182/blood-2022-169013)
- [Result] JX Yao, ARW O'Brien, YJ Tong*, Y Wang*. A Novel Finding in Cerebral Blood Flow in Patients with Sickle Cell Disease Using Bold Functional MRI. Blood (2022) 140 (Supplement 1): 5433-5434. (https://doi.org/10.1182/blood-2022-167594)
- [Result] SM Park, YY Ji, S Kwon, ARW O'Brien, Y Wang*, YL Kim*. Association of Noninvasive Peripheral Blood Hemoglobin Assessments with Venous Blood Draws Among Sickle Cell Patients. Blood (2022) 140 (Supplement 1): 7832-7833. (https://doi.org/10.1182/blood-2022-165132)
- See also: Indiana CTSI Study Listing — https://research-studies.allinforhealth.info/us/en/listing/11381/adultadultsteenteensteenagerteenagersadolescentadolescentssickle-cellsickle-cell-diseasepain-integrative-medicine-in-pain-management-in-sickle-cell-disease-assessing-the-clinical-efficacy-and-neurobiological-impact-with-acupuncture/